CLINICAL TRIAL: NCT05404074
Title: Pharmacokinetics of Cobitolimod Enemas in Participants With Active Ulcerative Colitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: InDex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSUC-02/21
Record Dates: First submitted 2022-05-17; First posted 2022-06-03 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — cobitolimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cobitolimod 500mg (Experimental): 2-3 single doses of rectal cobitolimod (500mg/50ml) over 3-6 weeks
  Interventions: Drug: Cobitolimod 500mg

INTERVENTIONS:
Drug: Cobitolimod 500mg — Rectal administration
  Other Names: Kappaproct

SUMMARY:
The purpose of the study is to evaluate the PK, safety and tolerability of cobitolimod ememas (500mg/50mL) given to participants with active left-sided UC.

DETAILED DESCRIPTION:
This is a single centre phase 1b study in participants with moderate to severe active UC designed to provide important supplementary data of the PK profile of cobitolimod.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Male or female participant aged ≥18 years.
3. Established diagnosis of UC, with minimum time from diagnosis of at least 3 months before screening.
4. Moderate to severe active left-sided UC (disease should extend 15 cm or more above the anal verge and may extend beyond the splenic flexure) determined by a 3-component Mayo score of 5 to 9 with an endoscopic subscore ≥2 (in sigmoid or descending segments) assessed by the Investigator's reading of the endoscopy, and with a stool frequency and rectal bleeding subscores each ≥1.
5. Clinically acceptable medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
6. Women only: WOCBP must practice abstinence (only allowed when this is the preferred and usual lifestyle of the participant) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]) from at least 4 weeks prior to dose to 4 weeks after last dose.

Women of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or females who have undergone hysterectomy or bilateral oophorectomy; or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] 25-140 IE/L is confirmatory)

Exclusion Criteria:

* 1. Suspicion of differential diagnosis such as Crohn's enterocolitis, ischaemic colitis, radiation colitis, indeterminate colitis, infectious colitis, diverticular disease, associated colitis, microscopic colitis, massive pseudopolyposis or non-passable stenosis.

  2. Acute fulminant UC, toxic megacolon and/or signs of systemic toxicity. 3. Have failed treatment with more than three advanced therapies (infliximab, adalimumab, golimumab, vedolizumab, ustekinumab or tofacitinib) of two different therapeutic classes (anti-TNF, anti-integrins, anti-IL12/23, JAK-inhibitors, or other approved advanced therapies for UC).

  4. Have had surgery for treatment of UC. 5. History of malignancy, unless treated with no relapse of the disease and ≥ 5 years since last treatment (cured) or treated (cured) basal cell or squamous cell in situ carcinoma.

  6. Serious known active infection e.g., any positive result on screening for serum hepatitis B surface antigen, hepatitis C virus antibodies and HIV.

  7. Gastrointestinal infections including positive Clostridium difficile stool assay (local laboratory reports must be available in accordance with normal clinic practice, to confirm that the current episode of disease exacerbation is not due to infection).

  8. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.

  9. Concomitant or planned treatment with cyclosporine, methotrexate, tacrolimus, or advanced therapies such as infliximab, adalimumab, golimumab, vedolizumab, ustekinumab or tofacitinib, or similar immunosuppressants and immunomodulators at enrolment. Any prior treatment with such drugs must have been discontinued at least 8 weeks prior to Visit 1 (except for ustekinumab, which must have been discontinued at least 12 weeks prior to Visit 1) or have non-measurable serum concentration levels.

  10. Treatment with rectal GCS, 5-ASA/SP or tacrolimus within 2 weeks before Visit 1.

  11. Long-term treatment (>14 days) with antibiotics or non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to Visit 1 (one short treatment regimen for antibiotics, occasional use of NSAIDs and low dose NSAIDs as prophylactic therapy is allowed).

  12. Females who are lactating or have a positive serum pregnancy test at Visit 1.

  13. Any planned major surgery within the duration of the study. 14. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1.

  15. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.

  16. Investigator considers the participant unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentrations (Cmax) | Week 6
  Maximum observed plasma concentrations (Cmax)
Time to Cmax (Tmax) | Week 6
  Time to Cmax (Tmax)
Area under the curve from 0 to timepoint t (AUCt) | week 6
  Area under the curve from 0 to timepoint t (AUCt)
AUC from 0 to infinity (AUCinf) | week 6
  AUC from 0 to infinity (AUCinf)
Half-life (T1/2) | week 6
  Half-life (T1/2)

SECONDARY OUTCOMES:
Frequency, intensity and seriousness of adverse events (AEs) | week 8
  Frequency, intensity and seriousness of adverse events (AEs)
Clinically significant changes in electrocardiogram (ECG), vital signs, safety laboratory | week 8
  Abnormal post-dose findings assessed by the Investigator as clinically significant will be reported as AEs.
Significant changes in blood biomarkers | week 8
  The difference between biomarker expression before and after treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Levin, Study Director — InDex Pharmaceuticals
Locations (1):
- CTC, Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No